CLINICAL TRIAL: NCT04025125
Title: Pathways to Cardiovascular Disease Prevention and Impact of Specialty Referral in Underrepresented Racial/Ethnic Minorities With HIV (Coordinating Center)
Brief Title: Pathways to Cardiovascular Disease Prevention (DCRI Central and Statistical Coordinating Center)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00101104; 1R01MD013493-01 (NIH)
Record Dates: First submitted 2019-07-02; First posted 2019-07-18 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS; Cardiovascular Diseases
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this research is to generate evidence-based recommendations for the management of cardiovascular disease (CVD) risk in People Living with HIV (PLWH). The overall objectives of this application are to demonstrate the effect of cardiology referral on CVD outcomes in a racially/ethnically diverse cohort of PLWH, and to generate qualitative data with which to develop of a future intervention. Our central hypothesis is that cardiology referral reduces incident CVD events in underrepresented racial/ethnic minority (URM) populations with HIV compared to nonreferral. Our hypothesis has been formulated based on our own work identifying that race and provider specialty impact cardiovascular risk management. The rationale for our research is that, once it is known how URM populations with HIV access cardiology referrals, and the impact on CVD outcomes, an intervention can be appropriately designed resulting in new and innovative approaches to the management of URM PLWH at elevated CVD risk.

DETAILED DESCRIPTION:
To identify factors associated with cardiology referral in under-represented racial and ethnic minority (URM) populations with HIV and elevated cardiovascular risk

ELIGIBILITY:
Project is not recruiting as retrospective review of electronic health records.

Inclusion Criteria:

Patient health records may be accessed from subjects who meet the following criteria:

1. Race equals Black/African-American, American Indian/Alaska Native, Asian, Native Hawaiian/Pacific Islander, or More than one race, and/or Ethnicity equals Hispanic or Latino;
2. Documented evidence of HIV positive status (HIV positive diagnosis (ICD10 codes B20-B24, or ICD9 codes 042, V08) and prescription of antiretroviral therapy (ART));
3. Documented evidence of elevated AtheroSclerotic CardioVascular Disease risk (ACC/AHA ASCVD 10 year risk ≥5%24, or Framingham Cardiovascular Disease 10 year risk ≥5%25) after HIV diagnosis. The date when the patient first meets either of these CVD risk thresholds and with 1 prior encounter not having CVD risk score defines the index time-point for Aim 1 of this study. These risk calculations depend on sex, age, body mass index, diabetes, current smoking, total cholesterol, HDL cholesterol, systolic blood pressure, and treatment for hypertension (defined from diagnosis codes). If cholesterol measures are not available, then body mass index may be used in place of lipids in the Framingham risk calculation; NOTE: must have a prior encounter within 365 days within health system prior to index
4. Presence of a modifiable risk factor: hypertension, diabetes, elevated total cholesterol, elevated LDL cholesterol and/or tobacco use.

Exclusion criteria:

1. Age <18 years of age or >99 years of age at index event;
2. Pre-existing ASCVD prior to index event, including a previous diagnosis of any acute myocardial infarction, heart failure, acute coronary syndromes, stable or unstable angina, arterial revascularization (includes coronary arterial or peripheral), stroke, transient ischemic attack or peripheral arterial disease presumed to be of atherosclerotic origin determined by ICD codes;
3. Encounter with cardiology specialist within 1 year prior to index
4. Evidence of ART for pre-exposure prophylaxis (i.e., Truvada [emtricitabine/tenofovir disoproxil fumarate] or post-exposure prophylaxis (e.g., Truvada plus raltegravir) without HIV diagnosis.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Project is not recruiting patients
  1. Race equals Black/African-American, American Indian/Alaska Native, Asian, Native Hawaiian/Pacific Islander, or More than one race, and/or Ethnicity equals Hispanic or Latino;
  2. Documented evidence of HIV positive status (HIV positive diagnosis and prescription of antiretroviral therapy (ART));
Sampling Method: Non-Probability Sample
Enrollment: 2039 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Bloomfield, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muiruri C, Corneli A, Cooper L, Dombeck C, Gray S, Longenecker CT, Meissner EG, Okeke NL, Pettit AC, Swezey T, Vicini J, Bloomfield GS. Perspectives of HIV specialists and cardiologists on the specialty referral process for people living with HIV: a qualitative descriptive study. BMC Health Serv Res. 2022 May 9;22(1):623. doi: 10.1186/s12913-022-08015-0. PMID 35534889
- [Result] Bloomfield GS, Hill CL, Chiswell K, Cooper L, Gray S, Longenecker CT, Louzao D, Marsolo K, Meissner EG, Morse CG, Muiruri C, Thomas KL, Velazquez EJ, Vicini J, Pettit AC, Sanders G, Okeke NL. Cardiology Encounters for Underrepresented Racial and Ethnic Groups with Human Immunodeficiency Virus and Borderline Cardiovascular Disease Risk. J Racial Ethn Health Disparities. 2024 Jun;11(3):1509-1519. doi: 10.1007/s40615-023-01627-0. Epub 2023 May 9. PMID 37160576
- [Result] Durstenfeld MS, Hill CL, Clare RM, Chiswell K, Sanders G, Gray S, Vicini J, Marsolo K, Okeke NL, Meissner EG, Thomas KL, Morse CG, Bloomfield GS, Pettit AC, Longenecker CT. Association of Cardiologist Clinic Visits With Cardiovascular Primary Prevention Outcomes Among People With HIV From Underrepresented Racial and Ethnic Groups in the Southern United States. J Am Heart Assoc. 2025 Mar 18;14(6):e038462. doi: 10.1161/JAHA.124.038462. Epub 2025 Mar 7. PMID 40055869
- [Result] Muiruri C, Dombeck C, Swezey T, Gonzales S, Lima M, Gray S, Vicini J, Pettit AC, Longenecker CT, Meissner EG, Okeke NL, Bloomfield GS, Corneli A. Specialty Care Referral for Underrepresented Minorities Living with HIV in the United States: Experiences, Barriers, and Facilitators. AIDS Patient Care STDS. 2024 Jun;38(6):259-266. doi: 10.1089/apc.2024.0066. Epub 2024 Jun 13. PMID 38868933

RESULTS

PARTICIPANT FLOW:
Recruitment Details: retrospective data study
Pre-assignment Details: As is pre-specified in the study protocol, Aim 3 data are not reported here.
Groups:
- Overall: cohort who have new elevated Cardiovascular Disease (CVD) risk
Period: Overall Study
Arm/Group | Overall
Started | 2039
Completed | 2039
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: Overall cohort.
Arm/Group | Overall
Number analyzed (Participants) | 2039
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45 [36 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1061
  Male | 978
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 225
  Not Hispanic or Latino | 1810
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9
  Asian | 35
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1755
  White | 65
  More than one race | 11
  Unknown or Not Reported | 164
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2039
Atherosclerotic Cardiovascular Disease (ASCVD) Risk Score [Median (Inter-Quartile Range); unit: 10-year risk percentage] — The ASCVD risk score is calculated using a formula developed by the American College of Cardiology (ACC) and the American Heart Association (AHA). The formula takes into account the individual's risk factors and outputs a 10-year risk percentage. The ASCVD risk score is categorized as follows: Low risk: < 5%, Borderline risk: 5-7.4%, Intermediate risk: 7.5-19.9%, High risk: ≥ 20%. Population: 1001 participants had data or were eligible for ASCVD analysis scoring.
  10-year risk percentage
    number analyzed (Participants) | 1001
    (all) | 5.1 [3.6 to 6.8]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Visit to a Cardiology Specialist From Cohort
Description: A binary variable, with 'yes' defined if there is documented evidence that a ambulatory visit was made with a cardiologist after becoming eligible by CVD risk score, and 'no' otherwise.
  Patients were followed from the date when they met eligibility criteria to the date of first encounter with a cardiology specialist or through a maximum of 5 years from their eligibility date. Follow-up was censored early at the end of data collection (December 31, 2020), or 6 months after the patient's last ambulatory visit, if earlier.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Overall: cohort who have new elevated CVD risk
Arm/Group | Overall
Number analyzed (Participants) | 2039
Participants | 283

2. Other Pre Specified Outcome: Incidence of All-cause Death
Description: Incidence of all-cause death will be determined from electronic health record data and a query of the National Death Index.
Time Frame: 5 years
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Incidence of Stroke
Description: Incidence of first stroke event will be determined from diagnosis and/or procedure codes from electronic health record data.
Time Frame: 5 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Incidence of Major Adverse Cardiovascular Event, Myocardial Infarction
Description: Incidence of first major adverse cardiovascular event (composite of cardiovascular death and myocardial infarction) will be determined from diagnosis and/or procedure codes from electronic health record data and a query of the National Death Index (Plus).
Time Frame: 5 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Provider Perspective on Facilitators and Barriers to Optimal CVD Prevention
Description: Qualitative information will be assessed from semi-structured interviews conducted with participating healthcare providers
Time Frame: Approximately 60 minutes
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Patient Perspective on Facilitators and Barriers to Optimal CVD Prevention
Description: Qualitative information will be assessed from semi-structured interviews conducted with participating patients
Time Frame: Approximately 60 minutes
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Proportion of Patients With Cholesterol Control
Description: Cholesterol control will be defined based on prevailing guidelines during the study period and will be evaluated based on cholesterol laboratory measures recorded in electronic health record data.
Time Frame: Longitudinal evaluation during 5 years of follow up.
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Proportion of Patients With Blood Pressure Control
Description: Blood pressure control will be defined based on prevailing guidelines during the study period (blood pressure <140/90 mmHg) and will be evaluated based on blood pressures recorded in electronic health record data.
Time Frame: Longitudinal evaluation during 5 years of follow up.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years
Description: This record is specific to Aim 1 only. Only all-cause mortality was collected.
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 137/2039
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT04025125/Prot_SAP_000.pdf